CLINICAL TRIAL: NCT01522963
Title: Medicinal Nicotine for Preventing Stress Induced Craving and Withdrawal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DA029689; R21DA029689 (NIH)
Record Dates: First submitted 2012-01-17; First posted 2012-02-01 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nicotine Lozenge Immediately Prior to Stress task (Experimental): Subjects will receive the nicotine lozenge immediately prior to the stress task at one laboratory session and after the stress task at the other laboratory session
  Interventions: Drug: Nicotine lozenge
- Nicotine lozenge 10 Minutes prior to Stress task (Experimental): Subjects will receive the nicotine lozenge after the stress task during one laboratory session and immediately prior to the stress task at the other laboratory session
  Interventions: Drug: Nicotine lozenge
- Nicotine lozenge 20 minutes prior to Stress task (Experimental): Subjects will receive the nicotine lozenge after the stress task during one laboratory session and 10 minutes prior to the stress task at the other laboratory session
  Interventions: Drug: Nicotine lozenge
- Nicotine Lozenge 30 minutes prior to stress taks (Experimental): Subjects will receive the nicotine lozenge 10 minutes prior to the stress task during one laboratory session and after the stress task at the other laboratory session
  Interventions: Drug: Nicotine lozenge

INTERVENTIONS:
Drug: Nicotine lozenge — A single dose of nicotine lozenge will be given at various timepoints relative to completion of a somewhat stressful task

SUMMARY:
The purpose of this study is to determine the timeframe (relative to a stress task) that is most effective at attenuating the increase in symptoms of tobacco craving and withdrawal that occur when smokers are presented with stressful situations.

ELIGIBILITY:
Inclusion Criteria:

* Smoking an average of at least 10 cigarette per day
* General good health

Exclusion Criteria:

* unstable medical or psychiatric conditions
* history of severe motion sickness
* women who are pregnant or breast feeding

The investigators will evaluate if there are other reasons why someone may not participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kotlyar, PharmD, Principal Investigator — University of Minnesota
Locations (1):
- Clinical and Translational Sciences Institute, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Kotlyar M, Lindgren BR, Vuchetich JP, Le C, Mills AM, Amiot E, Hatsukami DK. Timing of nicotine lozenge administration to minimize trigger induced craving and withdrawal symptoms. Addict Behav. 2017 Aug;71:18-24. doi: 10.1016/j.addbeh.2017.02.018. Epub 2017 Feb 10. PMID 28235705

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Lozenge Immediately Prior to Stress Task.: Subjects receive the 4 mg nicotine lozenge immediately prior to the stress task at one laboratory session and after the stress task at the other laboratory session
- Nicotine Lozenge 10 Min Prior to Stress Task: Subjects receive the 4 mg nicotine lozenge 10 minutes prior to the stress task at one laboratory session and after the stress task at the other laboratory session
- Nicotine Lozenge 20 Min Prior to Stress Task: Subjects receive the 4 mg nicotine lozenge 20 min prior to the stress task at one laboratory session and after the stress task at the other laboratory session
- Nicotine Lozenge 30 Min Prior to Stress Task: Subjects receive the 4 mg nicotine lozenge 30 min prior to the stress task at one laboratory session and after the stress task at the other laboratory session
Period: Overall Study
Arm/Group | Nicotine Lozenge Immediately Prior to Stress Task. | Nicotine Lozenge 10 Min Prior to Stress Task | Nicotine Lozenge 20 Min Prior to Stress Task | Nicotine Lozenge 30 Min Prior to Stress Task
Started | 24 | 25 | 25 | 24
Completed | 22 | 22 | 22 | 18
Not Completed | 2 | 3 | 3 | 6

BASELINE CHARACTERISTICS:
Population: Only those that completed the entire cross-over study were included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Lozenge Immediately Prior to Stress Task. | Nicotine Lozenge 10 Min Prior to Stress Task | Nicotine Lozenge 20 Min Prior to Stress Task | Nicotine Lozenge 30 Min Prior to Stress Task | Total
Number analyzed (Participants) | 22 | 22 | 22 | 18 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (10.6) | 39.7 (10.9) | 38.1 (16.2) | 37.9 (14.1) | 38.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 14 | 9 | 41
  Male | 14 | 12 | 8 | 9 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 1 | 3
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 8 | 4 | 1 | 20
  White | 14 | 11 | 16 | 14 | 55
  More than one race | 1 | 0 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 22 | 18 | 84

OUTCOME MEASURES:

1. Primary Outcome: Craving
Description: The difference between lozenge use at the designated time-point prior to the stress task and lozenge use after the stress task in craving response (measured by factor 1 of the Questionnaire on Smoking Urges) that occurs when smokers are exposed to a stressful task. The possible range of scores was between 5 and 35 with higher scores indicated greater smoking urges.
Time Frame: Baseline, 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nicotine Lozenge Immediately Prior to Stress Task. | Nicotine Lozenge 10 Min Prior to Stress Task | Nicotine Lozenge 20 Min Prior to Stress Task | Nicotine Lozenge 30 Min Prior to Stress Task
Number analyzed (Participants) | 22 | 22 | 22 | 18
units on a scale | 5.17 [2.43 to 7.91] | 2.45 [0.29 to 4.61] | -1.05 [-3.6 to 1.51] | -1.34 [-4.09 to 1.4]

2. Primary Outcome: Nicotine Withdrawal Symptoms
Description: The difference between lozenge use at the designated time-point prior to the stress task and lozenge use in withdrawal symptom response as measured by the Minnesota Nicotine Withdrawal Scale (MNWS) that occurs when smokers are exposed to a stressful task. The possible range of scores for the MNWS is between 0 and 28 with higher scores indicated greater withdrawal symptom severity.
Time Frame: 5 to 35 minutes
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nicotine Lozenge Immediately Prior to Stress Task. | Nicotine Lozenge 10 Min Prior to Stress Task | Nicotine Lozenge 20 Min Prior to Stress Task | Nicotine Lozenge 30 Min Prior to Stress Task
Number analyzed (Participants) | 22 | 22 | 22 | 18
units on a scale | 2.1 [0.23 to 3.98] | 2.18 [.07 to 4.29] | 0.32 [-1.88 to 2.51] | 0.16 [-1.95 to 2.28]

ADVERSE EVENTS:
Groups:
- Nicotine Lozenge Prior to Stress Task: Subjects will receive the nicotine lozenge at one of four time-points prior to the stress task at the first laboratory session and after the stress task at the second laboratory session
  Nicotine lozenge 4 mg: A single dose of nicotine lozenge will be given at various timepoints relative to completion of a somewhat stressful task
- Nicotine Lozenge After Stress Task: Subjects will receive the nicotine lozenge after the stress task during the first laboratory session and prior to the stress task at the second laboratory session
  Nicotine lozenge 4 mg: A single dose of nicotine lozenge will be given at various timepoints relative to completion of a somewhat stressful task
Arm/Group | Nicotine Lozenge Prior to Stress Task | Nicotine Lozenge After Stress Task
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/98
Other Adverse Events (participants affected / at risk) | 0/98 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No